CLINICAL TRIAL: NCT03884283
Title: A Post-market, Prospective, Multi-center, Nonrandomized Study to Assess Posterolateral Lumbar Fusions Using FIBERGRAFT BG Matrix
Brief Title: Prospective, Multi-center Study to Assess Posterolateral Fusion Using FIBERGRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prosidyan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CD0001
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Spinal Stenosis Lumbar
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: FIBERGRAFT BG Matrix — Subjects who meet the criteria for entrance into the study will undergo posterolateral fusion using FIBERGRAFT® BG Matrix in combination with autograft and bone marrow aspirate (BMA)

SUMMARY:
This is a prospective, non-randomized (single arm), multi-center, post-market clinical study designed to evaluate FIBERGRAFT® BG Matrix mixed with autograft and bone marrow aspirate in up to 150 subjects with degenerative disc disease (DDD) with or without radiculopathy, or spinal stenosis and/or spondylolisthesis requiring a fusion. The patient population will include adult (skeletally mature) men and women undergoing 1 or 2 level fusion in the lumbar spine (L2-S1) who are deemed eligible for the study, characterized by inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Is at least 18 years of age and skeletally mature.
3. Must have symptomatic spinal stenosis and/or spondylolisthesis or degenerative disc disease (DDD) at one or two adjacent levels from L2-S1, requiring a fusion.
4. Must have completed a minimum of three months of unsuccessful conservative, non-operative care.
5. DDD and spinal stenosis and/or spondylolisthesis must be confirmed by MRI or CT scans.
6. Must score at least 40 points on the Oswestry Disability Index.
7. Must score at least a 4 on a 10 cm Visual Analog Scale for back or leg pain.
8. Must be able to comply with the protocol's follow-up schedule.
9. Must understand and sign the IRB approved informed consent document.

Exclusion Criteria:

1. Symptomatic at more than two levels.
2. Previous fusion surgery at any lumbar level with or without instrumentation (prior discectomy, laminotomy, laminectomy or nucleolysis at the index level (> 6 months) is permitted).
3. Previous total disc replacement at any lumbar level.
4. Undergoing fusion for recurrent stenosis at the level to be treated.
5. Extraspinal cause of back and/or leg pain, or back and/or leg pain of unknown etiology.
6. Spondylolisthesis not able to be reduced to grade I.
7. Lumbar scoliosis greater than 11 degrees.
8. Osteoporosis*, osteopenia, osteomalacia, Paget's disease, or metabolic or systemic bone disorders that affect bone or wound healing.
9. Use of posterior instrumentation for stabilization is not possible.
10. Intra-operative soft tissue coverage is not possible.
11. Spinal tumors.
12. Active arachnoiditis.
13. Fractures of the epiphyseal plate or fractures for which stabilization of the fracture is not possible.
14. Impaired calcium metabolism.
15. Active systemic infection or surgical site infection.
16. Osteomyelitis at the graft site.
17. Rheumatoid arthritis or other autoimmune disease.
18. Chronic steroid use (used steroids for one month within the last 6 months) or any medical condition that requires treatment with drugs known to interfere with bone healing.
19. Systemic disease such as AIDS, HIV, hepatitis (active), tuberculosis.
20. Morbid obesity defined as body mass index (BMI) >40 or a weight more than 100 lbs over ideal body weight.
21. Smokers unless the subject agrees to quit at least 2 weeks prior to and for the duration of the study, confirmed by a carboxyhemoglobin test prior to surgery.
22. Psychosocial disorders that would preclude accurate evaluation or has a history of recent substance abuse.
23. Active malignancy except non-melanoma skin cancer; history of any invasive malignancy unless treated and in remission for at least five years.
24. Documented allergies to titanium.
25. Subjects with a history of anaphylaxis, history of multiple allergies, known allergies to bovine collagen, or who are being treated for desensitization to meat products because FIBERGRAFT® BG Matrix contains bovine collagen.
26. Pregnancy/able to become pregnant and not following a reliable contraceptive method, or interested in becoming pregnant in the next two years.
27. Participation in another investigational study within 30 days.
28. Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-05-21 (Actual)

PRIMARY OUTCOMES:
Spinal fusion | 12 months
  Spinal fusion will be determined via radiographic imaging at 12 months.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Long Beach Medical Center, Long Beach, California
  - Memorial Orthopaedic Surgical Group, Long Beach, California
  - Palm Beach Neurosurgery, Wellington, Florida
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Washington Spine & Scoliosis Institute at OrthoBethesda, Bethesda, Maryland
  - Northwell Health Orthopaedic Institute, Great Neck, New York
  - KeiperSpine, PC, Eugene, Oregon
  - Orthopedic and Neurologic Research Institute, Fort Worth, Texas
  - University of Virginia Orthopaedics, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided